CLINICAL TRIAL: NCT00005087
Title: Phase II Study of Paclitaxel and Cisplatin in Combination With Split Course Concomitant Hyperfractionated Re-Irradiation in Patients With Recurrent Squamous Cell Cancer of the Head and Neck
Brief Title: Paclitaxel, Cisplatin, and Filgrastim Combined With Radiation Therapy in Treating Patients With Locally Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9911; CDR0000067705
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Filgrastim; Cisplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation (BID) and chemotherapy (Experimental): Radiation (BID), cisplatin and paclitaxel given on days 1-5 (Monday-Friday) in weeks 1, 3, 5 and 7. G-CSF given on days 6-13.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel, cisplatin, and filgrastim combined with radiation therapy in treating patients who have locally recurrent head and neck cancer and have received previous treatment with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the median, one-year, and long-term (defined as two-year) disease-free survival and overall survival in patients with previously irradiated locally recurrent squamous cell cancer of the head and neck treated with paclitaxel, cisplatin, and filgrastim (G-CSF) combined with radiotherapy.
* Determine the rates of acute and late toxic effects of this regimen in these patients.
* Determine the pattern of disease progression in patients treated with this regimen.

OUTLINE: Patients undergo radiotherapy twice daily (4-6 hours apart) on days 1-5. Patients receive paclitaxel IV over 1 hour beginning immediately after completion of the first fraction of radiotherapy and completing less than 3 hours before starting the second fraction of radiotherapy on days 1-5. Patients receive cisplatin IV over 30 minutes beginning immediately after completion of paclitaxel infusion on days 1-5 and filgrastim (G-CSF) subcutaneously on days 6-13. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who initially respond to therapy but develop a recurrence with a resectable lesion (inside or outside the retreatment field) may undergo surgical resection.

Patients are followed at 4 weeks after completion of radiotherapy, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 34 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven locally recurrent primary squamous cell cancer (SCC) of the head and neck or second primary SCC of the head and neck

  * More than 1 prior recurrence allowed if the first recurrence occurred at least 6 months after completion of prior radiotherapy
* Disease must be confined to the head and neck (above the clavicles)
* No primary SCC of the nasopharynx or salivary gland
* Prior irradiation of 45-75 Gy to the majority (75% or greater) of tumor volume
* Entire tumor volume must be included in a treatment field that limits the total spinal cord dose (prior and anticipated) to 50 Gy

  * Prior radiotherapy records, including simulation and portal films, available in order to assure that cord tolerance is not exceeded
* Measurable disease
* Ineligible for complete surgical resection
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0 or 1

Life expectancy:

* No other concurrent illness that would limit survival

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Serum glutamate oxaloacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) no greater than 2 times normal*
* Alkaline phosphatase no greater than 2 times normal*
* * Greater than 2 times normal allowed if no metastases by liver ultrasound or CT scan

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* No other invasive malignancy within the past 2 years except in situ malignancies (e.g., carcinoma in situ of the cervix, carcinoma in situ of the breast, or nonmelanoma skin cancer)
* No other concurrent illness that would impair tolerance to therapy
* No grade 2 or worse pre-existing peripheral sensory neuropathy
* No hypersensitivity to E. coli derived products
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed as a component of the primary treatment
* No prior chemotherapy for recurrent disease
* At least 6 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 6 months since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2000-03; Primary Completion 2004-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From registration to 1 year

SECONDARY OUTCOMES:
Disease-free Survival | From registration to 1 year
Grade 4-5 toxicity | From one year after the start of radiation therapy to last follow-up.
Pattern of failure (local-regional, distant, new primary, death) | From registration to last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (235):
- United States (216):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Saint Agnes Cancer Center, Fresno, California
  - California Cancer Center, Fresno, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of St. Raphael, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Langer CJ, Harris J, Horwitz EM, Nicolaou N, Kies M, Curran W, Wong S, Ang K. Phase II study of low-dose paclitaxel and cisplatin in combination with split-course concomitant twice-daily reirradiation in recurrent squamous cell carcinoma of the head and neck: results of Radiation Therapy Oncology Group Protocol 9911. J Clin Oncol. 2007 Oct 20;25(30):4800-5. doi: 10.1200/JCO.2006.07.9194. PMID 17947728
- [Result] Horwitz EM, Harris J, Langer CJ, et al.: Concurrent split course hyperfractionated radiotherapy (Hfx RT), cisplatin (DDP) and paclitaxel (P) in patients with recurrent, previously irradiated squamous cell carcinoma of the head and neck (SCCHN): update of RTOG 9911 . [Abstract] J Clin Oncol 23 (Suppl 16): A-5577, 519s, 2005.
- [Result] Langer CJ, Harris J, Horwitz EM, Kies M, Ad VB, Wong SJ, Caudell JJ, Zeitzer KL, Spencer SA, Zhang Q, Yom SS, Le QT. Phase II Study of Low-Dose Paclitaxel and Cisplatin in Combination With Split-Course Concomitant Twice-Daily Reirradiation in Recurrent Squamous Cell Carcinoma of the Head and Neck: Long-term Follow-up of NRG Oncology RTOG 9911. Int J Radiat Oncol Biol Phys. 2026 Jan 1;124(1):50-60. doi: 10.1016/j.ijrobp.2025.07.1434. Epub 2025 Jul 31. PMID 40752652
- [Result] Langer CJ, Harris J, Horwitz E, et al.: Phase II trial of concurrent split course hyperfractionated radiotherapy (Hfx RT), cisplatin (DDP) and paclitaxel (P) in patients with recurrent, previously irradiated squamous cell carcinoma of the head and neck (SCCHN): results of RTOG 9911. [Abstract] J Clin Oncol 22 (Suppl 14): A-5509, 490s, 2004.